CLINICAL TRIAL: NCT03535064
Title: The Association of Hand Hygiene Practice on Primary Schoolgirls Absence Due to Upper Respiratory Infections (URIs) in Riyadh City, 2017-2018. A Cluster Randomized Trial
Brief Title: The Association of Hand Hygiene Practice on Primary Schoolgirls Absence Due to URIs in Riyadh City, 2017-2018.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abrar Alzaher (Other)
Responsible Party: Sponsor-Investigator, Abrar Alzaher, Principal Investigator, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-17-2523
Record Dates: First submitted 2018-05-12; First posted 2018-05-24 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Upper Respiratory Tract Infections
Keywords: HAND HYGIENE, HAND WASHING, INFLUENZA, SCHOOL ABSENCE, SCHOOL CHILDREN, UPPER RESPIRATORY INFECTIONS
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schools received hand hygiene workshop (Experimental): Schoolgirls of randomly assigned schools attended one-hour Arabic handwashing workshop conducted by the principal investigator one week after submitting all baseline questionnaires. Workshops included video-clip and interactive lecture about common infections in schools, methods of transmission, and hand washing procedure and time. Puzzle games related to hand hygiene were distributed among schoolgirls. Posters with cartoon princess picture promote for hand hygiene were also distributed among the schools.
  Interventions: Other: Hand Hygiene Workshop
- Schools with did not receive hand hygiene workshop (No Intervention): Schoolgirls in control group followed their usual hand washing procedure. When the study ended, schoolgirls of control school were exposed to the same intervention by the same investigator.

INTERVENTIONS:
Other: Hand Hygiene Workshop — Workshops included video-clip and interactive lecture about common infections in schools, methods of transmission, and hand washing procedure and time. Puzzle games related to hand hygiene were distributed among schoolgirls. Posters with cartoon princess picture promote for hand hygiene were also distributed among the schools.
  Arms: Schools received hand hygiene workshop

SUMMARY:
Research Problem:

Upper respiratory infections (URIs) are a common reason for absence from schools as it is estimated that children get six to eight episodes every year. In Jazan (2013-2014), 34% of primary health care centre attendees who were complaining of URIs were under 15 years old and 42% of them were positive when tested for viruses by nasopharyngeal swabs. An intervention for URIs prevention is hand hygiene, as it has been shown to have an impact on reducing the risk of respiratory infections by 50% among children in Karachi, Pakistan by encouraging hand washing with soap. Another randomised controlled trial study conducted in Spain among primary school students showed a statistically significant 38% reduction in the absenteeism rate due to URIs in the intervention group who received education about hand hygiene and used hand sanitisers which were distributed among schools. Also, the Chinese conducted a cluster randomised control trial evaluating the effect of a hand washing programme and revealed a 38% reduction in absence due to URIs among primary schoolchildren.

This preventive measure is questionable, as a randomised controlled trial done among primary school students in New Zealand revealed that encouraging the use of hand sanitisers in schools did not have an impact on reducing acute respiratory infections or absenteeism. The questionable effect was also documented in a systematic review and meta-analysis for randomised controlled trials about the effectiveness of hand hygiene in decreasing absences through illness in educational settings.

Research Significance:

Appropriate hand hygiene is recommended as a non-pharmacological preventive measure against respiratory infections. But this preventive measure is questionable as the results of randomised controlled trials about the effectiveness of different hand hygiene interventions in reducing absence due to upper respiratory tract infection in different educational settings are controversial. Furthermore, previous studies of hand hygiene interventions were low in quality and it is recommended to improve future studies relating to it. Also, there is no research on the effectiveness of these measures in Saudi Arabia. So, this piece will add new knowledge to local and international literature. In addition, this study may help the school health administration to develop a hand hygiene programme.

Objectives:

* To determine if hand hygiene education is associated with school absence rates due to URIs reduction among primary schoolgirls in Riyadh city, 2017-2018
* To measure post-intervention total primary schoolgirl's absence rate (both groups) in Riyadh city, 2017-2018.
* To measure post-intervention primary schoolgirls' absence rate due to upper respiratory infections (both groups) in Riyadh city, 2017-2018.

Methodology:

Cluster RCT will be conducted among primary schoolgirls attending public schools in Riyadh city in the first education semester. Sampling will be multistage to end up with four schools. 616 schoolgirls who are attending the selected classes will be invited to the study. Two schools will be randomly assigned to the intervention, which includes one-hour hand washing workshop at the beginning of the study, in addition to posters. Parents will self-administer the questionnaire at baseline, in addition to a follow-up phone interview questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All schoolgirls attended randomly selected schools

Exclusion Criteria:

* None

Ages: 6 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 496 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Primary schoolgirls absence due to URIs | five weeks
  Absence was collected from schools and parents were called to fill follow up questionnaire

SECONDARY OUTCOMES:
Total Primary schoolgirls absence | five weeks
  Absence was collected from schools

CONTACTS AND LOCATIONS:
Overall Officials: Abrar A Alzaher, MD, Principal Investigator — King Saud University
Locations (1):
- Ministry of Education, Riyadh, Saudi Arabia